CLINICAL TRIAL: NCT03626636
Title: A Randomized Controlled, Double-Masked, Crossover Clinical Trial Designed To Evaluate The Safety And Exploratory Efficacy Of 1.0 Mg Luminate® (Alg-1001) As A Treatment For Non-Exudative Macular Degeneration
Brief Title: A Clinical Trial Designed To Evaluate The Safety And Exploratory Efficacy Of 1.0 Mg Luminate® (Alg-1001) As A Treatment For Non-Exudative Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allegro Ophthalmics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Dry AMD
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Dry Age-related Macular Degeneration
MeSH Terms: interventions — risuteganib; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Treatment Group 1: 25 Non-Exudative AMD subjects with BCVA of 20/40 - 20/200 will be injected intravitreally with 1.0mg of Luminate®
  Interventions: Drug: Risuteganib
- Placebo Group (Placebo Comparator): Treatment Group 2: 15 Non-Exudative AMD subjects with BCVA of 20/40 - 20/200 will be treated with a sham injection
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Risuteganib — Subjects injected intravitreally with 1.0mg of Luminate®
  Other Names: ALG-1001, Luminate
  Arms: Active Group
Other: Sham — Sham injection
  Arms: Placebo Group

SUMMARY:
To evaluate the safety and exploratory efficacy of 1.0mg of Luminate® in patients with Intermediate Non-Exudative Macular Degeneration

DETAILED DESCRIPTION:
Approximately 40 eligible subjects who have been diagnosed with intermediate Non-Exudative AMD, that require treatment will be enrolled and randomized (1.7:1) to one of 2 treatment groups:

Treatment Group 1: 25 Non-Exudative AMD subjects with BCVA of 20/40 - 20/200 will be injected intravitreally with 1.0mg of Luminate® Treatment Group 2: 15 Non-Exudative AMD subjects with BCVA of 20/40 - 20/200 will be treated with a sham injection

At the 16-week visit, the study will be unmasked to the sponsor and injecting investigator (observing investigators will remain masked). Subjects in the treatment group will receive a 2nd dose of Luminate®. Subjects in the control group will be offered the opportunity to crossover to treatment with a single dose of Luminate®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 50 to 85 years of age at screening visit
* Subject has signed the Informed Consent form
* Subjects with Non-Exudative AMD having ETDRS BCVA between 33 and 72 letters read (equivalent to 20/40 - 20/200 on Snellen Chart) with the level of vision caused by the non-exudative AMD and no other factor/s
* Subjects with symptomatic decrease in visual acuity in the last 12 months
* Subjects with combination of areas of RPE disturbances (hyper or hypopigmentation) and/or > 1 large druse(n) (>125 microns) and/or multiple intermediate drusen (62-124 microns) in the macula as confirmed by the central reading center
* Subjects with evidence of reasonably well-preserved areas of RPE by clinical examination and well-defined RPE and outer segment ellipsoid line by OCT examination in the central 1 mm of the macula as confirmed by the central reading center. More specifically, reasonable reasonably well- preserved central 1 mm of the macula means:
* The RPE and outer retinal layers throughout the central 1 mm are intact
* No signs of NVAMD such as intraretinal or sub retinal fluid, or sub retinal hyper-reflective material
* No serous pigment epithelium detachments >100 microns in height

Exclusion Criteria:

* Females who are pregnant, nursing, planning a pregnancy during the study or who are of childbearing potential not using a reliable method of contraception and/or not willing to maintain a reliable method of contraception during their participation in the study. Women of childbearing potential with a positive urine pregnancy test administered at baseline are not eligible to receive study drug.
* Participation in an investigational drug or device study within 90 days of screening
* Subjects with active exudative AMD in the fellow eye
* Subjects who had anti-VEGF IVT in either eye in the past 90 days
* Subjects with pigment epithelium detachments
* Subjects with active exudative AMD
* Subjects with any prior retina surgery
* Subjects with pathology that could prevent observation and follow-up of macular structures and measurement of BCVA (i.e. advanced primary open angle glaucoma, any stage of normal tension glaucoma and corneal opacification)
* Subjects that are likely to require cataract surgery in the opinion of the investigator within the study protocol period

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Change in BCVA | 8 month total study including crossover
  1. Percentage of population with ≥ 8 letters (1 ½ lines) BCVA gain in the Luminate group (Treatment group 1 that received 2 doses of Luminate) from baseline to study week 28 vs the Sham control group from baseline to study week 12

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Derek Kunimoto, Gilbert, Arizona
  - Derek Kunimoto, Phoenix, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Raj Maturi, Indianapolis, Indiana
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lad EM, Boyer DS, Heier JS, Kornfield JA, Kuppermann BD, Quiroz-Mercado H, Aubel JM, Karageozian LS, Karageozian HL, Sarayba MA, Karageozian VH, Kaiser PK. Color Vision and Microperimetry Changes in Nonexudative Age-Related Macular Degeneration After Risuteganib Treatment: Exploratory Endpoints in a Multicenter Phase 2a Double-Masked, Randomized, Sham-Controlled, Crossover Clinical Trial. Ophthalmic Surg Lasers Imaging Retina. 2022 Aug;53(8):430-438. doi: 10.3928/23258160-20220725-02. Epub 2022 Aug 1. PMID 35951718
- [Derived] Boyer DS, Gonzalez VH, Kunimoto DY, Maturi RK, Roe RH, Singer MA, Xavier S, Kornfield JA, Kuppermann BD, Quiroz-Mercado H, Aubel J, Karageozian HL, Park JY, Karageozian VH, Karageozian L, Sarayba MA, Kaiser PK. Safety and Efficacy of Intravitreal Risuteganib for Non-Exudative AMD: A Multicenter, Phase 2a, Randomized, Clinical Trial. Ophthalmic Surg Lasers Imaging Retina. 2021 Jun;52(6):327-335. doi: 10.3928/23258160-20210528-05. Epub 2021 Jun 1. PMID 34185587

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03626636/Prot_SAP_000.pdf